CLINICAL TRIAL: NCT06303635
Title: Phase I Study to Evaluate the Safety and Immunogenicity of the Vaccine Booster With the Trivalent UFRJvac COVID-19 Vaccine
Brief Title: Safety of UFRJvac, Trivalent COVID-19 Vaccine
Acronym: UFRJvac-1
Status: Not yet recruiting | Type: Observational
Sponsor: Azidus Brasil (Industry)
Collaborators: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Sponsor
Other Study IDs: UFRJvac-1
Record Dates: First submitted 2024-03-08; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Healthy People
Keywords: UFRJvac

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Phase I study to evaluate the safety and immunogenicity of the vaccine booster with the trivalent UFRJvac COVID-19 vaccine.

DETAILED DESCRIPTION:
Phase I study to evaluate the safety and immunogenicity of the vaccine booster with the trivalent UFRJvac COVID-19 vaccine.

UFRJvac COVID-19 is a trivalent vaccine for preventing COVID-19. It is a protein subunit vaccine, being formulated with the entire recombinant spike protein ("S" protein, amino acids 1-1208) of the D614G, gamma and delta variants of SARS-CoV-2. One spike protein from each variant is expressed in HEK293 cells in trimeric form and stabilized in the prefusion conformation. In order for the adaptive immune response (humoral and cellular) to be enhanced against these proteins, the vaccine is formulated with the GLA-SE adjuvant.

The study will include 156 male or female participants aged between 18 and 65 years, with complete primary vaccination for COVID-19 and at least one booster dose, the last being carried out with the Comirnaty Bivalent BA.4/BA vaccine. 5.

UFRJvac COVID-19 will be administered once, as a booster dose, intramuscularly (0.5 mL), in doses of 5 μg or 15 μg of antigens.

Participants receive the investigational product on D0 and return for in-person medical evaluation on D2, D28, D84 and D168. Blood samples will be collected for humoral and cellular immunity tests on days D28, D84 and D168. On days D1, D3, D4, D5, D6 and D7 participants will be contacted by telephone to collect adverse events. Inclusion will be staggered, starting with 6 participants receiving PSI at a dose of 5 μg and distributed over at least 3 days. If tolerability is good, another 6 participants will receive the same dose and will also be distributed over at least 3 days. If tolerability is good, another 6 participants will receive the same dose and will be distributed over at least 3 days, totaling 18 participants with the lowest dose. If tolerability is good, another 18 participants receiving 15 μg will be included, also divided into 3 groups of 6 participants with at least 3 days of observation. If tolerability is good, an additional 120 participants will be included, 60 receiving the 5 μg dose and 60 receiving the 15 μg dose.

The main benefit of UFRJvac COVID-19 is to induce adaptive immunity against the three variants of SARS-CoV-2 (D614G, gamma and delta), and this combination of three antigens resulted, in preclinical studies, in a specific immune response also against the omicron variant. As this is a phase I study, there is still no data on adverse events related to the experimental drug. However, initially, reactions are expected at the site of product administration.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. Age from 18 to 65 years old, inclusive.
3. Complete primary vaccination for COVID-19 with one of the vaccines approved by ANVISA for use in Brazil, and at least one booster, the last of which must be with Comirnaty Bivalente BA.4/BA.5 between 4 and 18 months before vaccination. inclusion.
4. Body mass index (BMI) between 19.0 and 35.0 kg/m2, inclusive.
5. Female participant with a negative pregnancy test on the day of vaccination.
6. Consent form voluntarily signed before any procedure.

Exclusion Criteria:

1. Confirmation of active SARS-CoV-2 infection in rapid antigen test screening.
2. History of serious adverse reaction to any vaccine, medication or component of the investigational product.
3. History of immunodeficiency, autoimmune diseases and cardiomyopathies.
4. History of medium or major surgery within 3 months before inclusion.
5. History of malignancy within 1 year before screening (except basal cell carcinoma of the skin or in situ carcinoma of the cervix, which have already resolved).
6. History of uncontrolled coagulopathy or blood disorders that contraindicate intramuscular injection.
7. History of uncontrolled epilepsy or other progressive neurological disorders such as Guillain-Barré Syndrome.
8. Any decompensated chronic disease at the time of inclusion.
9. Treatment with immunosuppressive medications in the 3 months prior to the first vaccination or 6 months for chemotherapy.
10. History of systemic steroids (prednisone ≥ 20 mg/day or equivalent for >14 consecutive days) within 3 months prior to screening. Topical, inhaled, intranasal, and intra-articular corticosteroids are permitted regardless of dose.
11. Use of any other vaccine less than 14 days before or planning to use up to 29 days after V0.
12. Use of blood products in the 3 months before inclusion.
13. Use of another investigational product within 1 year before inclusion.
14. Pregnancy or breastfeeding at inclusion or planned during the study.
15. Fever or any acute illness within 1 week before inclusion. Participants who do not meet this criterion may be rescheduled for a new inclusion visit.
16. Presence of tattoos, scars, skin discoloration or any other skin disorders at the injection site that, in the opinion of the investigator, may impair the assessment of local reactogenicity.
17. Any condition that, in the opinion of the investigator, endangers the safety or rights of the participant or makes the participant unsuitable for the study.
18. Clinically significant changes in safety examinations, defined as:

    * Hb ≤ 10.9 g/dL;
    * Leukocyte count < 2500 cells/mm3;
    * Absolute neutrophil count < 1000 cells/mm3;
    * ESR outside normal values (18 to 65 years old, male - 2 to 28 mm; 18 to 65 years old, female - 2 to 36 mm);
    * ALT, AST and FA > 1.25 x ULN;
    * Total bilirubin > 1.1 x ULN;
    * Creatinine > 1.1 x ULN;
    * Glycated hemoglobin > 5.6%;
    * Troponin 1 > 0.16 ng/mL;
    * TP and aPTT > 1.1 x ULN;
    * CPK outside normal values (male adults - 38 to 174 U/L; female adults - 26 to 140 U/L);
    * C-reactive protein > 1.0 mg/dL.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include 156 male or female participants aged between 18 and 65 years, with complete primary vaccination for COVID-19 and at least one booster dose, the last being carried out with the Comirnaty Bivalent BA.4/BA vaccine. 5.
Sampling Method: Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2024-06-24 (Estimated); Primary Completion 2025-10-16 (Estimated); Study Completion 2025-11-25 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and reactogenicity of the UFRJvac COVID-19 vaccine booster | Up to 7 days after administration.
  Incidence, causality, severity and intensity of reported adverse events

SECONDARY OUTCOMES:
Evaluate the safety and reactogenicity of the vaccine booster with the trivalent UFRJvac COVID-19 | 28, 84 and 168 days after administration.
  Incidence, causality, severity and intensity of adverse events reported
Evaluate the humoral immunogenicity of the vaccine booster with the trivalent UFRJvac COVID-19 | 28, 84 and 168 days after vaccination.
  Increase in relation to the screening values of the geometric mean of the titer of neutralizing antibodies against the Wuhan and Ômicron variants of SARS-CoV-2
Evaluate the humoral immunogenicity of the vaccine booster the trivalent UFRJvac COVID-19 | 28, 84 and 168 days after vaccination.
  Percentage of participants with a 4-fold or greater increase from screening values in neutralizing antibody titers against the Wuhan and Omicron variants of SARS-CoV-2
Evaluate the humoral immunogenicity of the vaccine booster with the trivalent UFRJvac | 28, 84 and 168 days after vaccination.
  Increase in relation to the screening values of the geometric mean of the binding antibody (IgG) titer specific for protein S
Evaluate the humoral immunogenicity of the vaccine booster trivalent UFRJvac | 28, 84 and 168 days after vaccination.
  Percentage of participants with a 4-fold or greater increase from screening values in protein S-specific binding antibody (IgG) levels
Evaluate the cellular immunogenicity of the vaccine booster with the trivalent UFRJvac COVID-19 | 28, 84 and 168 days after vaccination.
  Increase over screening values in levels of IFN-γ, IL-2, TNF-α, IL4, IL5, and IL13 in culture supernatants from participant PBMCs

CONTACTS AND LOCATIONS:
Overall Officials: Jose Cerbino Neto, MD, Principal Investigator — Instituto D'Or de Ensino e Pesquisa

IPD SHARING:
Plan to Share IPD: No